CLINICAL TRIAL: NCT00128895
Title: Prevention of Relapses in PR3-ANCA-associated Vasculitis, a Tailored Approach
Brief Title: Prevention of Relapses in Proteinase 3 (PR3)-Anti-neutrophil Cytoplasmic Antibodies (ANCA)-Associated Vasculitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Arthritis Association (Industry); Dutch Kidney Foundation (Other)
Responsible Party: Principal Investigator, J.S.F. Sanders, dr JSF Sanders, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZA-ANCA-1
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Vasculitis
Keywords: Wegener's granulomatosis, ANCA, vasculitis, proteinase 3; ANCA-associated vasculitis; ANCA
MeSH Terms: conditions — Vasculitis; Granulomatosis with Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- azathioprine, standard (Active Comparator): standard azathioprine maintenance upto one year after diagnosis, subsequently tapering of azathioprine with 25 mg per 3 months
  Interventions: Drug: azathioprine
- azathioprine, longterm (Experimental): longterm maintenance with azathioprine upto four years after diagnosis, subsequently azathioprine will be tapered with 25 mg per 3 months
  Interventions: Drug: azathioprine

INTERVENTIONS:
Drug: azathioprine — azathioprine 2 mg/kg oral once daily, duration according to arm

SUMMARY:
Treatment of patients with PR3-ANCA-associated vasculitis consists of two phases: remission induction with highly effective, but also relatively toxic, drugs and, secondly, after remission is achieved, maintenance therapy with less toxic drugs. Currently, remission-maintenance therapy with azathioprine is stopped after approximately 18 months. However, the optimal duration of azathioprine maintenance therapy is unknown.

The investigators have found that patients with PR3-ANCA-associated vasculitis who remain cytoplasmic anti-neutrophil cytoplasmic autoantibody (C-ANCA) positive after induction of remission have an increased risk to experience relapse of disease. Therefore they will test whether relapse risk in these patients can be reduced by extending maintenance therapy at the cost of acceptable therapy related toxicity. After induction of stable remission, ANCA will be measured by immunofluorescence (IIF). C-ANCA positive patients will be randomized for either standard therapy with azathioprine (until 18 months after diagnosis), or longterm azathioprine maintenance therapy (until 48 months after diagnosis).

DETAILED DESCRIPTION:
Treatment of patients with PR3-ANCA-associated vasculitis consists of two phases: remission induction with highly effective, but also relatively toxic, drugs and, secondly, after remission is achieved, maintenance therapy with less toxic drugs. Currently, remission-maintenance therapy with azathioprine is stopped after approximately 18 months. However, the optimal duration of azathioprine maintenance therapy is unknown.

The investigators have found that patients with PR3-ANCA-associated vasculitis who remain C-ANCA positive after induction of remission have an increased risk to experience relapse of disease (MC Slot et al. Arthritis Rheum. 2004 15;51(2):269-73). Therefore they will test whether relapse risk in these patients can be reduced by extending maintenance therapy at the cost of acceptable therapy related toxicity. After induction of stable remission, ANCA will be measured by IIF. C-ANCA positive patients will be randomized for either standard therapy with azathioprine (until 18 months after diagnosis), or longterm azathioprine maintenance therapy (until 48 months after diagnosis).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ANCA-associated vasculitis
* PR3-ANCA antibodies present
* Indication for treatment with cyclophosphamide and prednisolone

Exclusion Criteria:

* Intolerance or allergy to azathioprine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2003-06; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
disease free survival | four years after diagnosis

SECONDARY OUTCOMES:
cumulative organ damage | four years after diagnosis
side-effects | up to four years after diagnosis
cumulative dosages of cyclophosphamide, prednisolone and azathioprine | up to four years after diagnosis
quality of life | four years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Coen A Stegeman, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (8):
- Netherlands (8):
  - VU University Medical Centre, Amsterdam
  - University Medical Centre Groningen, Groningen
  - Martini Hospital Groningen, Groningen
  - Medical Centre Leeuwarden, Leeuwarden
  - University Hospital Maastricht, Maastricht
  - UMC St Radboud, Nijmegen
  - Erasmus Medical Centre, Rotterdam
  - University Medical Centre Utrecht, Utrecht

REFERENCES:
- [Result] Sanders JS, de Joode AA, DeSevaux RG, Broekroelofs J, Voskuyl AE, van Paassen P, Kallenberg CG, Tervaert JW, Stegeman CA. Extended versus standard azathioprine maintenance therapy in newly diagnosed proteinase-3 anti-neutrophil cytoplasmic antibody-associated vasculitis patients who remain cytoplasmic anti-neutrophil cytoplasmic antibody-positive after induction of remission: a randomized clinical trial. Nephrol Dial Transplant. 2016 Sep;31(9):1453-9. doi: 10.1093/ndt/gfw211. Epub 2016 May 30. PMID 27242368